CLINICAL TRIAL: NCT00410982
Title: Gemcitabine Combined With Busulfan and Melphalan, With Hematopoietic Cell Transplantation, for Patients With Poor-prognosis Advanced Lymphoid Malignancies
Brief Title: Gemcitabine Plus Busulfan, Melphalan and Hematopoietic Cell Transplant for Advanced Lymphoid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0803
Record Dates: First submitted 2006-12-11; First posted 2006-12-13 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2012-09

CONDITIONS: Leukemia; Lymphoma; Myeloma
Keywords: Lymphoid Malignancies; Hodgkin's Disease; Non-Hodgkin's Lymphoma; Acute Lymphoblastic Leukemia; Chronic Lymphocytic Leukemia; Hematopoietic Cell Transplantation; Myeloma; Leukemia; Lymphoma; Busulfan; Busulfex; Myleran; Gemcitabine; Gemcitabine Hydrochloride; Gemzar; Melphalan; Alkeran
MeSH Terms: conditions — Leukemia; Lymphoma; Neoplasms, Plasma Cell; Hodgkin Disease; Lymphoma, Non-Hodgkin; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Busulfan; Gemcitabine; Melphalan; Stem Cell Transplantation; Rituximab; Fibroblast Growth Factor 7

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine + Busulfan + Melphalan + HCT (Experimental): HCT = Hematopoietic Cell Transplantation
  Interventions: Drug: Busulfan; Drug: Gemcitabine; Drug: Melphalan; Other: Hematopoietic Cell Transplantation; Drug: Rituximab for Patients with B-Cell Malignancies; Drug: Palifermin

INTERVENTIONS:
Drug: Busulfan — Day -10 = 32 mg/m^2 Intravenous Test Dose; Days -8 thru -5 = 105 mg/m^2 Intravenous
  Other Names: Busulfex; Myleran
Drug: Gemcitabine — Day -8 = 75 mg/m^2 Intravenous bolus; Day -3 = 75 mg/m^2 Intravenous bolus.
  Other Names: Gemzar; Gemcitabine Hydrochloride
Drug: Melphalan — Day -3 and Day -2 = 60 mg/m^2 Intravenous.
  Other Names: Alkeran
Other: Hematopoietic Cell Transplantation — Infusion of stem cells on Day 0.
  Other Names: Stem Cell Infusion; HCT
Drug: Rituximab for Patients with B-Cell Malignancies — 375 mg/m^2 Intravenous on Days 1 and 8.
  Other Names: Rituxan
Drug: Palifermin — 60 microgram/kg by vein on Days -13 to -11 and Days 0, +1, +2
  Other Names: Kepivance

SUMMARY:
The goal of this clinical research study is to find the highest tolerated dose of gemcitabine that can be given with busulfan and melphalan. The safety of this drug combination will also be studied.

DETAILED DESCRIPTION:
Busulfan and melphalan are designed to kill cancer cells by binding to DNA (the genetic material of cells), which may cause cancer cells to die. They are commonly used in stem cell transplantation.

Gemcitabine is designed to disrupt the growth of cancer cells, which may cause cancer cells to die. It may help to increase the effect of busulfan and melphalan on the tumor cells, by not allowing these cells to repair the DNA damage caused by busulfan or melphalan.

You will have apheresis done to collect some of your stem cells. Apheresis is the process of removing part of the blood (such as platelets or white blood cells) from the body in order to remove certain elements, such as stem cells. Then, the rest of the blood is returned back to your body. Your stem cells will be put back in your body after you finish receiving gemcitabine, busulfan, and melphalan. Apheresis will be done by a major vein through a central venous catheter (CVC), usually in the chest. A CVC is a sterile flexible tube that will be placed into a large vein while you are under local anesthesia. Your doctor will explain these procedures to you in more detail, and you will be required to sign a separate consent form for each procedure.

If you are found to be eligible to take part in this study, you will be enrolled in a group of at least 2 participants to begin receiving the study drugs. The dose of the study drugs you receive will depend on when you enrolled in this study. If no intolerable side effects occur in your group, researchers will continue to enroll participants at the next highest dose level until the highest tolerable dose of the study drugs is found. The dose that you receive will remain the same throughout this study.

Before you start to receive chemotherapy at treatment doses, you will be given a very small test dose of busulfan. Blood (1 teaspoon) will be drawn to check the levels of the drug in your blood at ten different timepoints (5-6 tablespoons total). This will help the study staff calculate your treatment doses of this drug. If there is a schedule conflict and the laboratory is not available for this testing, this procedure will not be performed. In that case, you would receive an unchanging dose of busulfan during the treatment.

During Day 1 you will receive gemcitabine and busulfan by CVC.

On Days 2-4, you will receive busulfan.

On Day 5, you will not receive any study drugs.

On Day 6, you will receive gemcitabine followed by melphalan.

On Day 7, you will receive melphalan.

On Day 8, you will not receive any study drugs.

On Day 9, you will receive your autologous stem cells through a needle in your vein over about 30-60 minutes.

If you have a B-cell cancer, you will receive rituximab (a treatment used for certain lymphomas or chronic lymphocytic leukemia) as part of standard of care, 1 day after and again 8 days after the infusion of the autologous cells.

As part of standard care, you will receive G-CSF (filgrastim) as an injection just under your skin daily, starting 1 day after the transplant, until your blood cell levels return to normal.

As part of standard care, you will receive a total of 6 doses of palifermin by vein. Three (3) of the doses will be given before starting chemotherapy (with a 24-hour break between the last dose of palifermin and the first dose of chemotherapy), and 3 doses will be given after the last chemotherapy dose, starting on Day 0.

You will be taken off this study 100 days after the transplant. You may be taken off this study early if the disease gets worse or you experience any intolerable side effects.

As part of standard care, you will remain in the hospital for about 3-4 weeks after transplantation. After you are released from the hospital, you will continue as an outpatient in the Houston area to be monitored for infections and transplant-related complications.

This is an investigational study. Busulfan, gemcitabine, and melphalan are all FDA approved and commercially available. The use of these study drugs together and the use of gemcitabine at these dose levels is investigational. Up to 143 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - <70 years.
2. Patients with lymphoid malignancies who do not qualify for treatment protocols of higher priority: 2.1) Primary refractory/recurrent Hodgkin's disease 2.2) Primary refractory/recurrent non-Hodgkin's lymphoma 2.3) Multiple myeloma beyond first remission or unresponsive to therapy, who do not qualify for higher priority melphalan-based protocols.
3. Adequate renal function, as defined by estimated serum creatinine clearance >/= 50 ml/min and/or serum creatinine </= 1.8 mg/dL.
4. Adequate hepatic function, as defined by Serum glutamic oxaloacetic transaminase (SGOT) and/or serum glutamic-pyruvic transaminase (SGPT) </= 3 * upper limit of normal; serum bilirubin and alkaline phosphatase </= 2 * upper limit of normal.
5. Adequate pulmonary function with forced expiratory volume for 1 second (FEV1), forced vital capacity (FVC) and Carbon Monoxide Diffusing Capacity (DLCO) >/= 50% of expected corrected for hemoglobin or volume.
6. Adequate cardiac function with left ventricular ejection fraction >/= 40%. No uncontrolled arrhythmias or symptomatic cardiac disease.
7. Zubrod performance status <2.
8. Patient should be willing to participate in the study by providing written consent.
9. Negative Beta HCG text in a woman with child-bearing potential, defined as not post-menopausal for 12 months or no previous surgical sterilization

Exclusion Criteria:

1. Patients with grade >/= 3 non-hematologic toxicity from previous therapy that has not resolved to grade 1.
2. Patients with prior whole brain irradiation
3. Patients with active hepatitis B virus (HBV), either active carrier (HBsAg +) or viremic (HBV DNA >=10,000 copies/mL, or >= 2,000 IU/mL).
4. Evidence of either cirrhosis or stage 3-4 liver fibrosis in patients with chronic hepatitis C or positive hepatitis C serology.
5. Active infection requiring parenteral antibiotics.
6. Human immunodeficiency virus (HIV) infection, unless the patient is receiving effective antiretroviral therapy with undetectable viral load and normal CD4 counts
7. Patients having received radiation therapy to head and neck (excluding eyes), and internal organs of chest, abdomen or pelvis in the month prior to enrollment.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2006-12; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Gemcitabine with Busulfan + Melphalan | Baseline to Day 100 post transplant, up to 115 days
  MTD defined as dose level where one of two participants enrolled at a given time have no dose limiting toxcities (DLT) at that dose level. Continual reassessment from baseline for DLT, monitored daily during hospitalization, weekly to Day 30 and monthly to Day 100. Dose level assessed with each 21-day dose escalation cycle, Gemcitabine delivered Day -8 to Day -5 of 21 day cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Yago Nieto, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Nieto Y, Gruschkus S, Valdez BC, Jones RB, Anderlini P, Hosing C, Popat U, Qazilbash M, Kebriaei P, Alousi A, Saini N, Srour S, Rezvani K, Ramdial J, Barnett M, Gulbis A, Shigle TL, Ahmed S, Iyer S, Lee H, Nair R, Parmar S, Steiner R, Dabaja B, Pinnix C, Gunther J, Cuglievan B, Mahadeo K, Khazal S, Chuang H, Champlin R, Shpall EJ, Andersson BS. Improved outcomes of high-risk relapsed Hodgkin lymphoma patients after high-dose chemotherapy: a 15-year analysis. Haematologica. 2022 Apr 1;107(4):899-908. doi: 10.3324/haematol.2021.278311. PMID 33951890
- See also: The University of Texas MD Anderson Cancer Center official website — http://www.mdanderson.org